CLINICAL TRIAL: NCT02486549
Title: A Prospective Randomized Comparison of Ultrasound-guided Supraclavicular and Interscalene Block in Patients Undergoing Arthroscopic Shoulder Surgery
Brief Title: Supraclavicular Versus Interscalene Block for Shoulder Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tokat Gaziosmanpasa University (Other)
Responsible Party: Principal Investigator, Tuğba Karaman, Assistant Professor, M.D., Tokat Gaziosmanpasa University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: artroscopy
Record Dates: First submitted 2015-06-24; First posted 2015-07-01 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Pain
Keywords: Pain; Anesthesia Recovery Period; Brachial Plexus
MeSH Terms: conditions — Pain | interventions — Bupivacaine; Ultrasonography

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Supraclavicular Block (Experimental): Ultrasound guided supraclavicular block with 20 ml of 0.25% bupivacaine will be performed
  Interventions: Procedure: Supraclavicular Block; Drug: Bupivacaine; Device: Ultrasound
- Interscalene block (Active Comparator): Ultrasound guided inter scalene block with 20ml of 0.25% bupivacaine will be performed.
  Interventions: Procedure: Interscalene Block; Drug: Bupivacaine; Device: Ultrasound

INTERVENTIONS:
Procedure: Supraclavicular Block — Under ultrasound guidance an insulated needle is advanced with in- plane technique into the brachial plexus sheath and 20ml 0.25% bupivacaine will be administered
  Arms: Supraclavicular Block
Procedure: Interscalene Block — Under ultrasound guidance an insulated needle will be placed through the middle scalene muscle,into the interscalene groove with in-plane technique and 20ml 0.25%bupivacaine will be administered into the brachial plexus
  Arms: Interscalene block
Drug: Bupivacaine — 20ml 0.25% bupivacaine will be injected for brachial plexus block
  Other Names: Marcaine
Device: Ultrasound — The Ultrasound will be used for brachial plexus visualization

SUMMARY:
The purpose of this study is to compare the supraclavicular block to interscalene block in patients undergoing arthroscopic shoulder surgery.

DETAILED DESCRIPTION:
The aim of this study is to evaluate the efficacy of the supraclavicular block in comparison with interscalene block on postoperative pain, quality of recovery and side effects in patients undergoing arthroscopic shoulder surgery under general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing shoulder surgery in American Society of Anesthesiologists physical status I-II

Exclusion Criteria:

* with a known allergy to study medications,
* chronic opioid use,
* ipsilateral upper limb neurological deficits,
* severe respiratory disease,
* coagulopathy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Postoperative Pain | up to postoperative 24 hours
  The visual analog scale will be used for assessment

SECONDARY OUTCOMES:
Quality of recovery | in the postoperative 24 hours
  The Quality of Recovery-40 (QR40) questionnaire will be used for assessment
Motor block | up to postoperative 24 hours
  The muscle force will be evaluated with scale 0 to 3( 0:normal muscle force, 1: reduced muscle force, 2: impaired mobility 3: paralysis
Sensory block | up to postoperative 24 hours
  The sensorial block will be assessed by pinprick test.
Adverse events | up to postoperative 24 hours
  The number of patients with adverse events will be recorded.
Analgesics requirement time | up to postoperative 24 hours
  the first intravenous analgesic requirement time will be recorded.
Systolic Blood pressure changes | at time of surgery
  The blood pressure will be measured non invasively and the systolic blood pressure lower than 90 mmHg or decrease more than 20% of baseline will be accepted as a hypotension.
Heart rate changes | at time of surgery
  The heart rate will be assessed via electrocardiographic monitoring and recorded as beat/minute.

CONTACTS AND LOCATIONS:
Overall Officials: Tugba Karamanaraman, M.D., Principal Investigator — Gaziosmanpasa University Medical School
Locations (1):
- Gaziosmanpasa University Medical School, Tokat Province, Turkey (Türkiye)